CLINICAL TRIAL: NCT05135923
Title: The Effect of Gluten-free Diet on Gut Microbiota and Metabolic Regulation in People With Coeliac Disease
Brief Title: Glutenfree, Gut Microbiota and Metabolic Regulation
Acronym: GRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other); Det Glutenfrie Verksted (Unknown)
Responsible Party: Principal Investigator, Vibeke Telle-Hansen, Associate professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20/02822
Record Dates: First submitted 2021-10-12; First posted 2021-11-26 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Random Allocation; Double-Blind Method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benchmark gluten-free products (Active Comparator): Products containing less than 6g fibre per 100g product.
  Interventions: Dietary Supplement: Randomized, controlled trial (RCT) with parallel arms and double blinded
- Optimised gluten-free products (Experimental): Products containing less than 6g fibre per 100g product.
  Interventions: Dietary Supplement: Randomized, controlled trial (RCT) with parallel arms and double blinded

INTERVENTIONS:
Dietary Supplement: Randomized, controlled trial (RCT) with parallel arms and double blinded — Experiment group receive optimized gluten free products (high in fiber and whole grain) compared to comparable benchmark gluten free products (control group).

SUMMARY:
High intake of dietary fiber provides health benefits and reduces the risk of developing cardio-metabolic diseases, such as type 2 diabetes (T2D) and cardiovascular disease (CVD). The intake of fiber is below the recommendations worldwide. In Norway, bread and cereals represent a major source of fiber. A low fiber intake is evident for people with celiac disease due to the removal of wheat, rye and barley from the diet. We therefore need to increase our knowledge in relation to fiber-rich food that will be tolerated also by people with celiac disease. The aim of the study is to investigate the effect of fiber rich gluten free products on blood glucose levels compared to benchmark gluten free products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with celiac disease
* BMI 18.5-27
* 18-65 years

Exclusion Criteria:

* chronic metabolic diseases, such as diabetes (type 1 and 2), cardiovascular diseases, cancer the last six months
* gut diseases, including chron's disease, ulcerative colite
* food allergies or intolerance, except for coliac disease
* pregnant and/or lactating
* smokers
* BMI <18.5 and >27
* planned weight reduction and/or 5% weight change the last three months
* blood donor the last two months and during the study period
* not willing to stop using dietary supplements, including probiotic products, cod liver oil etc, four weeks before and throughout the study
* use of antibiotics < three months before study start and throughout the study period
* alcohol consume > 40 g/day
* hormone treatment (except for contraceptives)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration of blood glucose | 3 weeks
  Blood analyses of glucose (fasting and post-prandial (after an OGTT)) before and after intervention with benchmark versus optimized gluten-free products.

SECONDARY OUTCOMES:
Concentration of blood cholesterol, triglycerides, fatty acids, C-peptide | 3 weeks
  Blood analyses of total cholesterol, triglycerides, fatty acids, and C-peptide (fasting) before and after intervention with benchmark versus optimized gluten-free products.
Concentration of blood inflammatory markers | 3 weeks
  Blood analyses of inflammatory markers (fasting) before and after intervention with benchmark versus optimized gluten-free products.
Feces microbiota analyses performed with Bio-Me's Precision Microbiome Profiling platform (PMP) | 3 weeks
  Feces analyses of microbiota before and after intervention with benchmark versus optimized gluten-free products.
Gastrointestinal Symptoms Rating Scale-Irritable bowl syndrome (GSRS-IBS) | 3 weeks
  GSRS-IBS analyses before and after intervention with benchmark versus optimized gluten-free products with the following response scale: 1 (no discomfort at all) to 7 (very severe discomfort)
Concentration of satiety hormones in blood | 3 weeks
  Blood analyses of satiety hormones (fasting) before and after intervention with benchmark versus optimized gluten-free products.
Bristol Stool Chart (BSC) | 3 weeks
  BSC analyses before and after intervention with benchmark versus optimized gluten-free products with a scale from 1 (separate hard lumps, like nuts) to 7 (watery, no solid pieces).

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo Metropolitan University, Oslo, Norway